CLINICAL TRIAL: NCT02948543
Title: Adding Mitomycin to Bacillus of Calmette-Guerin (BCG) as Adjuvant Intravesical Therapy for High-risk, Non-Muscle-invasive Bladder Cancer: a Randomised Phase 3 Trial
Brief Title: Adding Mitomycin to BCG as Adjuvant Intravesical Therapy for High-risk Non-Muscle-invasive Bladder Cancer
Acronym: BCG+MM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Cancer Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1301; 12613000513718 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2016-08-01; First posted 2016-10-28 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; BCG Connaught; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Arm B):Intravesical BCG + MM (Experimental): Induction (weekly x 9); and followed by Maintenance (monthly x 9) beginning 3 months after randomisation.
  Dosage of Bacillus of Calmette-Guerin (BCG) dependent on preferred brand of BCG by participating institution. Either 2-8 x 10^8 CFU for OncoTICE or, 81mg for ImmuCYST and TheraCys. Prior to treatment commencement, investigators should nominate which BCG brand will be used. The same brand of BCG must be used for all treatment administered to an individual participant throughout the study.
  Dosage of Mitomycin (MM) fixed at 40mg per instillation.
  Interventions: Biological: Bacillus of Calmette-Guerin (BCG); Drug: Mitomycin (MM)
- Treatment (Arm A): Intravesical BCG (Other): Induction (weekly x 6); and followed by Maintenance (monthly x 10) beginning 3 months after randomisation.
  Dosage of Bacillus of Calmette-Guerin (BCG) dependent on preferred brand of BCG by participating institution. Either 2-8 x 10^8 CFU for OncoTICE or, 81mg for ImmuCYST and TheraCys. Prior to treatment commencement, investigators should nominate which BCG brand will be used. The same brand of BCG must be used for all treatment administered to an individual participant throughout the study.
  Interventions: Biological: Bacillus of Calmette-Guerin (BCG)

INTERVENTIONS:
Biological: Bacillus of Calmette-Guerin (BCG) — A strain of tubercle bacillus which modifies biologic response.
  Other Names: OncoTICE; ImmuCYST; TheraCys
Drug: Mitomycin (MM) — An antibiotic produced by a soil actinomycete which inhibits DNA synthesis.
  Arms: Treatment (Arm B):Intravesical BCG + MM

SUMMARY:
Open label, randomised phase 3 trial of the addition of Mitomycin to BCG as adjuvant intravesical therapy for high-risk, non-muscle-invasive bladder cancer. The study aim is to compare disease-free survival between treatment arms: BCG alone versus Mitomycin in addition to BCG.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

Background:

Instillation of Bacillus of Calmette-Guerin (BCG) into the urinary bladder (intravesical administration) improves rates of disease recurrence and progression after transurethral resection (TUR) of high risk, non-muscle-invasive bladder cancer (NMIBC), but over 30% of people still develop recurrent transitional cell carcinoma (TCC) despite optimal therapy with adjuvant intravesical BCG. Our meta-analysis, including a recent randomised phase 2 trial, suggests that outcomes might be improved further by using an adjuvant intravesical regimen that includes both Mitomycin (MM) and BCG. These promising findings require corroboration in a definitive, large scale, randomised phase 3 trial using standard techniques for intravesical administration.

General Aim:

To determine the efficacy and safety of MM in addition to BCG in patients with NMIBC.

Design:

Open label, randomised, stratified, 2-arm multicentre phase 3 clinical trial. Population: The target population is adults with resected, high-risk NMIBC (high grade Ta or any grade T1) suitable for intravesical chemotherapy treatment. Key eligibility criteria include: prior transurethral resection of all visible tumour, adequate organ function, and ECOG performance status 0-2.

Study Treatments:

Arm A: Intravesical BCG Alone (standard): Induction (weekly x 6), followed by Maintenance (monthly x 10); or Arm B: Intravesical BCG + MM (experimental): Induction (weekly x 9), followed by Maintenance (monthly x 9).

Statistical Considerations:

A sample size of 500 (followed until 213 events are observed) provides 85% power to detect a 10% improvement in disease free survival (DFS) rate at 2 years from 70% on BCG alone to 80% on BCG and MM (hazard ratio 0.63) at a significance level of 0.05, allowing for 10% non-compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with confirmed high grade pTa or stage pT1 (any grade) non-muscle invasive bladder cancer on initial or re-resection histology (concurrent carcinoma in situ is allowed).
2. Age >= 18 yrs
3. No macroscopically visible disease at cystoscopy within 8 weeks prior to randomisation. This may be either the initial Transurethral Resection of the Bladder Tumour (TURBT) at which the primary tumour was completely resected, or a planned second cystoscopy and/or re-resection done within 8 weeks of the initial TURBT.
4. ECOG Performance Status of 0-2
5. Adequate bone marrow, renal and liver function confirmed by pre-randomisation blood tests.
6. Study treatment both planned and able to start within 4 weeks of randomisation
7. Has completed the HRQL questionnaires or is unable to complete them because of literacy, insufficient English or limited vision
8. Willing and able to comply with all study requirements, including treatment, timing and/or nature of all required assessments
9. Signed, written informed consent

Exclusion Criteria:

1. Contraindications or hypersensitivity to investigational products, BCG and Mitomycin
2. Prior treatment with any other intravesical agent including BCG or Mitomycin (excludes single doses given post TURBT)
3. Current or past transitional cell carcinoma (TCC) of the upper urinary tract
4. Prior muscle-invasive (stage T2 or higher) transitional-cell carcinoma of the bladder
5. Bladder dysfunction precluding intravesical therapy eg. Severe urinary incontinence or overactive or spastic bladder
6. Life expectancy < 3 months
7. Congenital or acquired immune deficiencies, whether due to a concurrent disease (e.g. acquired immune deficiency syndrome (AIDS), leukaemia, lymphoma) or immunosuppressive therapy (e.g. corticosteroids), or cancer therapy (cytotoxic drugs, radiation)
8. Prior radiotherapy of the pelvis
9. Prior or current treatment with radiotherapy-response or biological-response modifiers
10. Clinical evidence of existing active tuberculosis
11. History of another malignancy within 5 years prior to registration. Patients with non-melanomatous carcinoma of the skin are eligible for this study.
12. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol.
13. Pregnancy, lactation, or inadequate contraception. Women must be post menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilised or use a (double if required) barrier method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2013-07; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (death or recurrence) | Up to 5 years
  Measured from the date of randomisation until the date of disease recurrence, upper tract disease is first evident, or the date of death, or until the date last known to be alive and without disease recurrence. Assessed via cystoscopy.

SECONDARY OUTCOMES:
Activity (Clear cystoscopy at 3 months) | At 3 months after patient randomised
  Treatment activity is defined as a negative cystoscopy & biopsy at nominal week 12 (i.e. after induction therapy, but prior to the commencement of maintenance therapy). Assessed via cystoscopy and biopsy.
Time to recurrence (recurrence) | Up to 5 years
  Measured from the date of randomisation until the first date recurrence is detected. Disease recurrence is defined as evidence on cystoscopy or biopsy of Ta or T1-4 disease, or if there is evidence of metastatic disease. Assessed via cystoscopy.
Time to progression (disease progression) | Up to 5 years
  Measured from the date of randomisation until the first date progression is detected. Disease progression is defined as evidence of disease that is of a higher grade or a higher stage than at baseline. Assessed via cystoscopy.
Safety (Adverse events graded according to CTC AE V4.0) | Measured before day 1 of each instillation during treatment.
  The NCI Common Terminology Criteria for Adverse Events version 4 (NCI CTCAE v4.03) will be used to classify and grade the intensity of adverse events after each treatment cycle.
Health-Related Quality of Life | Up to 5 years from the date of randomisation
  Health related quality life is a composite outcome aggregated to arrive at one reported value to ensure multiple aspects of the participants life are adequately assessed and measured. The following questionnaires will be used; the 24-item EORTC Bladder Symptoms Quality of Life module (QLM-BLS24); the EORTC Core Quality of Life Questionnaire (QLQ-C30); and the International Prostate Symptom Score (I-PSS).
Overall survival time (death from any cause) | Up to 5 years
  Overall survival is defined as the interval from the date of randomisation to the date of death from any cause or the date last known to be alive.
Treatment Completion | Measured at end of study treatment (12 months after patient randomized).
  Treatment completion is defined as having received 75% or more of the planned numbers of induction and maintenance doses.
Marginal resource use | 5 years after last patient randomized (or date last patient has died, whichever sooner).
  Assessed via a specifically designed resource utilisation form (collecting information such as number, type and duration of visits).

OTHER OUTCOMES:
Exploratory Tissue Biomarker Investigation | Baseline
  Optional donation of formalin-fixed paraffin embedded (FFPE) tumour tissue for future biological or translational sub-studies. These future studies may include investigations of how BCG + MM may work in people with Non-Muscle-invasive Bladder Cancer as well as studies that may help to understand the pathogenic course of this cancer and related diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Dickon Hayne, Study Chair — Fiona Stanley Hospital
Locations (17):
- Australia (16):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Southside Cancer Care Centre, Miranda, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - GenesisCare, St Leonards, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland
  - Footscray Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Austin Health - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital - City Campus, Parkville, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Nottingham City Hospital - City Campus, Nottingham, United Kingdom